Stadistical analysis plan

## Online Training Program on Social Cognition for Patients With Schizophrenia

NCT ID not yet assigned

ULaguna 18-12-2019

## Study title: TRAINING IN COGNITION AND SOCIAL COMPETENCE IN PATIENTS WITH SCHIZOPHRENIA

A single-blind randomized clinical trial will be carried out in patients suffering from schizophrenia and who have the legal capacity to consent to the study. Study participants will be randomized to either the experimental group (e-Motional Training) plus Individual Placement and Support (IPS) or the control group (IPS alone).

For data analysis, taking into account that not all patients will have pre and post information, general mixed models will be used with identification of the subject and repeated time measurements (pre and post).

It will be carried out for the analysis of the mean tests as variance (t-student test of independent samples and Levene's test of equality of variances),

The efficacy of a training program in cognition and social competence (e-Motional Training) will be evaluated in patients with schizophrenia when improving the recognition of basic emotions, social cognition, emotional intelligence and social competence.

## INFORMATION ON THE USE OF RESOURCES AND FUNDING

## (mandatory compliance)

| Do you need funding for this study? | YES | | NO | ) X |
|---|---|---|---|---|
| Do you have required funding for this study? | YES X NO | | ) | |
| How many hours of your time during work hours will you dedicate to | 25% | | | |
| this study? | | | | |
| Do you have the material means (equipment, techniques, others? | YES | X | NO | ) |
| Where will the study take place? | | | | |
| CONSULTING DAY UICEC HOSPITALIZATION | X | OTHE | RS | SINPROMI |
| ROOM HOSPITAL | | | | |
| Will additional tests be performed outside of routine clinical practice?* | YES | | NO | ) X |
| *If YES, indicate below: | | | | |
| Use of biological samples: | YES | | NO | ) X |
| *If YES, indicate their location below: | | | | |
| SERVICE / DEPARTMENT: PSYCHIATRY SERVICE. ULL. | | | | |
| COLLECTION | YES | | NO | ) X |
| BIOBANK | YES | | NO | ) X |
| Use of patient clinical data: | | | | |
| Transfer of encrypted data (pseudonymized) outside the EU to the | YES | | NO | ) X |
| entities of our group, to service providers or to scientific researchers | | | | |
| who collaborate with us | | | | |